CLINICAL TRIAL: NCT05056714
Title: Development of a Severity Assessment Score for Nasosinus Polyposis (PSI Score)
Acronym: PSI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: PSI
Record Dates: First submitted 2021-09-16; First posted 2021-09-24 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2023-02

CONDITIONS: Nasal Polyposis
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Nasosinus Polyposis: patients with Nasosinus Polyposis included in the study
  Interventions: Other: Questionaries

INTERVENTIONS:
Other: Questionaries — The patient will answer several questionaries

SUMMARY:
nasosinus polyposis (=PNS) is a chronic inflammatory disease of the nasal cavity and sinus cavity with a prevalence of 2 to 4% in the general population. The functional impact of PNS has a major impact on one's quality of life.Medical treatment, nasal irrigations and local glucocorticoids as well as short treatment of oral glucocorticoids have shown a short-term benefit versus placebo. Surgery improves the efficacy of local treatments, but 40% of patients have a recurrence of polyps at 18 months and 20% of patients require a surgery recovery at 5 years. The development of monoclonal antibodies directly targeting the inflammatory way is a real public health issue. Bachert C. et al recently demonstrated the efficacy of Dupilumab (anti-IL-4/13 antibody) injected subcutaneously on the overall symptomatology of PNS. The marketing authorization (AMM) for the first biotherapy to be available soon includes PNS's severe nature and resistance to treatment, although there is no consensus definition or score to characterize this severity. This study aims at developping a score for assessing severity in PNS. We suggest that this assessment strategy could be applied to the PNS. The originality and the innovative character of this project is the statistical modeling behind the creation of the score. Thus, the importance of symptoms, anatomical and biological factors, the estimation of the quality of life of the patients, the level of care use and the number of surgeries all become measurable indicators that are a direct reflexion of the severity and the control of PNS, called latent variables because they cannot be directly measured. To consider this detail, modeling using structural equations seems optimal to develop a severity score (PSI score) of PNS in order to personalize the therapeutic care of patients. Main Objective: To develop a severity score for PNS using latent variable modeling: Polyps Severity Index (PSI)

DETAILED DESCRIPTION:
In practice, during their otolaryngologist (ORL) consultation, patients will have a complete clinical check-up and will be prescribed the necessary complementary examinations if they have not already been performed recently (<6 months). All data will be collected in an anonymous database.

The patient will answer a questionnaire to evaluate the cardinal symptoms of PNS using a visual scale from 0 to 10. He will then have a standard ORL clinical check-up (otoscopy, then rhinoscopy with speculum and nasal endoscopy) in order to make a nasal anatomical assessment (duration 5 minutes).

They will be given a questionnaire on admission to the waiting room to find out the impact of their nasal discomfort on their quality of life (score used routinely and validated in the literature, SNOT-22), as well as a questionnaire concerning their asthma if it exists (score used routinely and validated in the literature, ACT). The importance of the endoscopic involvement will be evaluated using the Lidholt score (see Appendix) and the importance of the radiological involvement directly from the CT or Cone beam computed tomography (=CBCT) results using the Lund-MacKay score. The estimated time to complete these questionnaires and to assess the endoscopic and radiological involvement is an additional 10 minutes. Blood will be drawn (as part of the initial routine workup) to assess complete blood count (for blood hypereosinophilia) and IgE levels (serum and total IgE). We will repeat the assessment routinely performed as part of the follow-up of patients with PNS by questionnaire, interview and physical check-up at 3 months when the patients return for their follow-up visit. No additional exams or questionnaires to the routine workup will be performed for this study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Patients included are all adult (>18 years) patients with PNS: Inflammation of the nose and sinuses that is characterised by two or more of the following symptoms (at least one of which must be nasal obstruction or runny nose):
* Nasal obstruction and nasal congestion
* Rhinorrhoea (anterior or posterior)
* Facial pain or pressure
* Decreased or loss of sense of smell
* Sneezing and/or nasal pruritus

These symptoms should be associated with :

* Endoscopic signs of nasal polyps
* Diffuse bilateral naso-sinusal opacities on CT or CBCT

Exclusion Criteria:

* Decline to participate in the study
* No one who speaks or understands French
* History of skull base surgery for tumours
* History of major head trauma
* History of cerebral-facial radiotherapy or chemotherapy
* History of inflammatory or neurodegenerative neurological pathology
* Systemic disease associated with the presence of sinus polyps (Granulomatosis - with polyangiitis, cystic fibrosis, primary ciliary dyskinesia, immune deficiency)
* Cancer or haematological disease in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nasosinisal polyposis identified or followed up
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Develop a severity score for PNS using latent variable modeling: Polyps Severity Index (PSI) | 3 months
  the estimated value of the structural coefficients relating measurable indicators of PNS to the endogenous latent variable: the severity of the disease (PSI score).

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Hôpital kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHU Liile, Lille
  - Hôpital de la Croix Rousse, Lyon
  - CHU Lyon Sud, Lyon
  - Hôpitaux Universitaires de Marseille Conception, Marseille
  - Hôpital Lariboisiere, Paris

IPD SHARING:
Plan to Share IPD: No